CLINICAL TRIAL: NCT02841995
Title: A Phase 2a, Dose-Escalation, Open-Label Study to Evaluate the Safety, Tolerability, and Activity of KD025 in Subjects With Chronic Graft Versus Host Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Activity of KD025 in Subjects With Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT17631; KD025-208 (Other: Kadmon)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Graft vs Host Disease
Keywords: cGVHD; Allogeneic hematopoietic stem cell transplantation; Immune System Diseases; Steroid refractory chronic graft vs host disease (cGVHD); Bone Marrow Transplantation; Anti-Inflammatory Agents; Glucocorticoids; Corticosteroids
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases | interventions — belumosudil; KD025

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Belumosudil 200 mg QD (Experimental): Participants received belumosudil 200 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 64.2 months).
  Interventions: Drug: Belumosudil (KD025)
- Cohort 2: Belumosudil 200 mg BID (Experimental): Participants received belumosudil 200 mg orally BID in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 45.9 months).
  Interventions: Drug: Belumosudil (KD025)
- Cohort 3: Belumosudil 400 mg QD (Experimental): Participants received belumosudil 400 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 49.2 months).
  Interventions: Drug: Belumosudil (KD025)

INTERVENTIONS:
Drug: Belumosudil (KD025) — Pharmaceutical form: Capsules or Tablets Route of administration: Oral
  Other Names: SLx-2119; REZUROCK

SUMMARY:
This study was been conducted to evaluate the safety, tolerability, and activity of belumosudil (formerly known as KD025) in adult participants with chronic graft versus host disease (cGVHD).

DETAILED DESCRIPTION:
Fifty four (54) participants were enrolled to receive orally administered belumosudil 200 milligrams (mg) once daily (QD), belumosudil 200 mg twice daily (BID), or belumosudil 400 mg QD.

Study drug was administered in 28-day cycles until disease progression or occurrence of unacceptable toxicity. Participants received study drug in the inpatient or outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female participants at least 18 years of age who had allogenic bone marrow transplant (BMT) or hematopoietic stem cell transplantation (HSCT).
* Received glucocorticoid therapy and calcineurin therapy or glucocorticoid therapy alone for cGVHD at study entry. Participants on calcineurin therapy only, without glucocorticoid therapy, were not eligible. Participants also received other therapies thought not to be immunosuppressive (such as extracorporeal photopheresis; ECP), were considered for enrollment in this study on a case-by-case basis.
* Had persistent active cGVHD manifestations, as defined by 2014 NIH Consensus Development Project on Criteria for Clinical trials in cGVHD, after at least 2 months of steroid therapy.
* No more than 3 prior lines of treatment for cGVHD.
* Karnofsky Performance Scale of greater than (>) 40.
* Adequate organ and bone marrow functions evaluated during the 14 days prior to enrollment as follows:

  * Absolute neutrophil count greater than or equal to (>=) 1.5*10^9/L (without myeloid growth factors within 1 week of study entry)
  * Platelet count >=50*10^9/L (without transfusion or thrombopoietin or thrombopoietin analogues within 2 weeks of study entry)
* Adequate safety laboratory values:

  * Total bilirubin less than or equal to (<=) 1.5*upper limit of normal (ULN)
  * Alanine aminotransferase and aspartate aminotransferase <=3*ULN
  * Glomerular filtration rate (GFR) >= 30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) using the 4-Variable Modification of Diet in Renal Disease variable formula
* Female participants of childbearing potential have a negative pregnancy test at screening. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had any evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, anti estrogens, or ovarian suppression.
* Women of childbearing potential (i.e., menstruating women) must had a negative urine pregnancy test (positive urine tests were to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.
* Sexually active women of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes:

  * Intrauterine device plus one barrier method;
  * Stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method;
  * 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or
  * A vasectomized partner
* For male participants who were sexually active and who were partners of premenopausal women: agreement to use two forms of contraception as in criterion 10 above during the treatment period and for at least 3 months after the last dose of study drug.
* Able to provide written informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* Female participant who was pregnant or breastfeeding.
* Received an investigational GVHD treatment within 28 days of study entry.
* Had acute GVHD.
* Taken any medication known to be a moderate or strong inhibitor of the cytochrome (CY) CYP3A4 isozyme or any drugs that are moderate or strong CYP3A4 inducers.
* History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease or coronary artery disease).
* Regular and excessive use of alcohol within the 6 months prior to study entry defined as alcohol intake >14 drinks per week in a man or >7 drinks per week in a woman. Approximately 10 grams of alcohol equals one "drink" unit. One unit equals 1 ounce of distilled spirits, one 12-ounce beer, or one 4-ounce glass of wine.
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years of enrollment, with the exception of completely resected basal cell or squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low-risk prostate cancer after curative resection.
* Relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
* Had previous exposure to belumosudil or known allergy/sensitivity to belumosudil or any other Rho-associated protein kinase-2 inhibitor.
* Taken other immunosuppressant drugs for GVHD, including mammalian target of rapamycin inhibitors (Note: Only steroids, calcineurin inhibitors, and ECP are acceptable).
* Corrected QT interval using Fridericia's formula >450 milliseconds.
* Female participant who was pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of Minnesota, Minneapolis, Minnesota
  - Oncology Hematology Care, Cincinnati, Ohio
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SJ, Cutler C, Blazar BR, Tu A, Yang Z, Pavletic SZ. Correlation of Patient-Reported Outcomes with Clinical Organ Responses: Data from the Belumosudil Chronic Graft-versus-Host Disease Studies. Transplant Cell Ther. 2022 Oct;28(10):700.e1-700.e6. doi: 10.1016/j.jtct.2022.06.020. Epub 2022 Jul 1. PMID 35781099
- [Derived] Jagasia M, Lazaryan A, Bachier CR, Salhotra A, Weisdorf DJ, Zoghi B, Essell J, Green L, Schueller O, Patel J, Zanin-Zhorov A, Weiss JM, Yang Z, Eiznhamer D, Aggarwal SK, Blazar BR, Lee SJ. ROCK2 Inhibition With Belumosudil (KD025) for the Treatment of Chronic Graft-Versus-Host Disease. J Clin Oncol. 2021 Jun 10;39(17):1888-1898. doi: 10.1200/JCO.20.02754. Epub 2021 Apr 20. PMID 33877856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 active sites in the United States. A total of 64 participants were screened between 15 September 2016 and 08 March 2018, of which 10 participants were screen failures due to not meeting eligibility criteria.
Pre-assignment Details: A total of 54 participants were enrolled and treated with belumosudil in the study.
Groups:
- Cohort 1: Belumosudil 200 mg QD: Participants received belumosudil 200 milligrams (mg) orally once daily (QD) in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 64.2 months).
- Cohort 2: Belumosudil 200 mg BID: Participants received belumosudil 200 mg orally twice daily (BID) in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 45.9 months).
Period: Overall Study
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Started | 17 | 16 | 21
Completed | 0 | 0 | 0
Not Completed | 17 | 16 | 21
Not completed — Disease progression | 5 | 11 | 8
Not completed — Withdrawal by Subject | 2 | 4 | 4
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Investigator decision | 2 | 0 | 1
Not completed — Death | 0 | 0 | 2
Not completed — Noncompliance to protocol | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 0 | 0
Not completed — Other | 4 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD | Total
Number analyzed (Participants) | 17 | 16 | 21 | 54
Age, Continuous [Median (Full Range); unit: years] | 50.0 [20 to 63] | 55.0 [30 to 75] | 46.0 [25 to 75] | 51.5 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 9 | 20
  Male | 13 | 9 | 12 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 15 | 14 | 19 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response (OR)
Description: OR was defined as the percentage of participants with complete response (CR) or partial response (PR). The OR determination of chronic graft versus host disease (cGVHD) was based on cGVHD response assessment performed by clinicians as per the 2014 National Institutes of Health (NIH) Consensus Development Project for Clinical Trials in cGVHD criteria. CR was defined as the resolution of all manifestations in each organ or site. PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site; and cGVHD progression was defined as the clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.
Time Frame: From the date of randomization to the date of first documentation of progression or death due to any cause or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
percentage of participants | 64.7 [38.3 to 85.8] | 68.8 [41.3 to 89.0] | 57.1 [34.0 to 78.2]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (defined as the time from the first dose of study drug up to 28 days after the last dose of study drug). TEAEs included both SAEs and non-SAEs.
Time Frame: From first dose of study drug up to 28 days after the last dose of study drug (maximum duration: up to 64.2 months)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Participants
  TEAE | 17 | 16 | 20
  TESAE | 5 | 6 | 13

3. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR was defined as the participants with either a CR or PR or lack of response (LOR), where LOR included the response status of unchanged (LOR-U), mixed (LOR-M), or progression (LOR-P). BOR was assessed per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria. CR was defined as the resolution of all manifestations in each organ or site; PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site; LOR-M was defined as CR or PR in at least one organ accompanied by progression in another organ, LOR-U was defined as outcomes that did not meet the criteria for CR, PR, progression or mixed response, LOR-P was defined as progression in at least one organ or site without a response in any other organ or site.
Time Frame: as for outcome 1
Population: Analysis was performed on mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Participants
  CR | 0 | 0 | 0
  PR | 11 | 11 | 12
  LOR-U | 2 | 3 | 4
  LOR-M | 2 | 1 | 0
  LOR-P | 2 | 1 | 1

4. Secondary Outcome: Number of Participants With Maximal Improvement From Baseline in Global Severity Rating (GSR) by Clinician-reported cGVHD Assessment
Description: The GSR assessment was performed by asking the participants to rate their disease severity of cGVHD symptoms on a 0 to 10-point numeric rating scale, where score 0 indicated 'not at all severe cGVHD symptoms' and score 10 indicated 'most severe cGVHD symptoms possible'. The response was defined using scores from 9 organs: skin, eyes, mouth, esophagus, upper gastrointestinal (GI) track, lower GI tract, liver, lungs, and joints and fascia plus GSR. End of treatment (EOT) visit was performed within 3 days after participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. Maximal improvement from Baseline was calculated as lowest GSR score on scheduled visits minus GSR score at Baseline with possible ranges from -10 to 10. The lower the number means the better improvement in cGVHD symptoms. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Baseline up to end of treatment (i.e., up to 64.2 months)
Population: Analysis was performed on mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Participants
  -7 | 0 | 0 | 2
  -6 | 0 | 2 | 0
  -5 | 2 | 2 | 0
  -4 | 2 | 0 | 3
  -3 | 4 | 0 | 1
  -2 | 2 | 4 | 4
  -1 | 1 | 2 | 4
  0 | 5 | 4 | 3
  1 | 0 | 1 | 1
  3 | 0 | 1 | 0
  Missing | 1 | 0 | 3

5. Secondary Outcome: Number of Participants With Maximal Improvement From Baseline in Symptom Activity by cGVHD Activity Assessment Participant Self-Report
Description: cGVHD symptom severity was self-reported by participants. Participants were asked to rate their disease symptom severity over the last week on the following questions: skin itching at its worst, moth dryness at its worst, mouth pain at its worst, mouth sensitivity at its worst, main compliant on eyes, symptom severity on eyes. Severity rating was done on a 0 to 10-point numeric rating scare, where score 0 indicated 'not at all severe cGVHD symptoms' and score 10 indicated 'most severe cGVHD symptoms possible'. EOT visit was performed within 3 days after participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. Maximal improvement from Baseline was calculated as the lowest symptom severity score on scheduled visits minus the symptom severity score at Baseline with possible ranges from -10 to 10. The lower the number means the better improvement in cGVHD symptoms.
Time Frame: From Baseline up to end of treatment (i.e., up to 64.2 months)
Population: Analysis was performed on mITT population. Only those categories in which at least 1 participant had data were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Participants
  -8 | 0 | 0 | 1
  -7 | 3 | 2 | 0
  -6 | 0 | 1 | 4
  -5 | 2 | 0 | 2
  -4 | 2 | 2 | 1
  -3 | 2 | 2 | 2
  -2 | 2 | 3 | 2
  -1 | 2 | 2 | 2
  0 | 1 | 1 | 0
  1 | 0 | 0 | 1
  2 | 0 | 1 | 2
  4 | 1 | 0 | 0
  Missing | 2 | 2 | 4

6. Secondary Outcome: Failure-free Survival (FFS)
Description: Failure-free survival was defined as the time (in months) from first dose of study drug to either the start of another new systemic treatment for cGVHD, relapse of the underlying disease or death. If no such events happened, FFS was censored by last response assessment or long term follow up assessment, whichever was the latest and available. Kaplan-Meier survival method was used for the analysis.
Time Frame: From first dose of study drug to either start of another new systemic treatment for cGVHD, relapse of the underlying disease or death or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
months | 10.6 [3.78 to NA] — 95% confidence interval (CI) upper limit was not available because of the less number of participants with event. | 9.8 [4.01 to 19.02] | 9.7 [2.60 to 16.10]

7. Secondary Outcome: Change From Baseline in Corticosteroids Dose
Description: Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline up to end of treatment (i.e., anytime up to 64.2 months)
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per kilogram per day
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 15 | 19
milligrams per kilogram per day | -0.110 (0.101) | -0.111 (0.147) | -0.116 (0.152)

8. Secondary Outcome: Number of Participants With Change From Baseline in Calcineurin Inhibitor (CNI) Usage
Description: Calcineurin inhibitors included systemic tacrolimus and cyclosporine. Number of participants who took CNI at Baseline and had reduction and discontinuation in CNI use as compared to Baseline during the study are reported in this outcome measure. EOT visit was performed within 3 days after the participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication.
Time Frame: Baseline up to end of treatment (i.e., anytime up to 64.2 months)
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants who had taken CNI at Baseline and with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 6 | 6 | 11
Participants
  Participants with reduction in CNI dose | 5 | 5 | 6
  Participants who discontinued CNI | 0 | 1 | 3

9. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time (in weeks) from first documentation of response to the time of first documentation of deterioration from best response (e.g., CR to PR, or PR to LR). LOR included the response status of unchanged (LOR-U), mixed (LOR-M), or progression (LOR-P). Per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site; PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site; LOR-M was defined as CR or PR in at least one organ accompanied by progression in another organ, LOR-U was defined as outcomes that did not meet the criteria for CR, PR, progression or mixed response, LOR-P was defined as progression in at least one organ or site without a response in any other organ or site. Kaplan-Meier was used for the analysis.
Time Frame: From the date of first response until documented disease progression or death due to any cause or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on responder population which included participants who received at least 1 dose of study medication and achieved a PR or CR response at any post-baseline response assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 11 | 11 | 12
weeks | 40.0 [8.14 to NA] — 95% CI upper limit was not available because of the less number of participants with event. | 10.9 [2.00 to 35.14] | 15.9 [4.14 to 38.14]

10. Secondary Outcome: Time-to-Response (TTR)
Description: Time-to-response was measured as the time (in weeks) from first dose of study drug to the time of first documentation of response. Response was defined as the participants achieving a PR or CR at any post-baseline response assessment. Per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site and PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: From first dose of study drug treatment to the time of first documentation of response or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on responder population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 11 | 11 | 12
weeks | 8.14 [7.9 to 26.1] | 8.14 [4.1 to 40.0] | 8.07 [4.1 to 67.0]

11. Secondary Outcome: Percentage of Participants With Best Response in Each Individual Organ
Description: Best response was defined as the percentage of participants with CR or PR. Response was assessed per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site; PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site. Organ response assessment was performed on 9 individual organs: skin, eyes, mouth, esophagus, upper gastrointestinal (GI), lower GI, liver, lungs, and joints and fascia and is reported in this outcome measure.
Time Frame: From date of randomization until disease progression or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category. Here, '0' in the number analyzed field signifies that none of the participants were available for the analysis at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
percentage of participants
  Skin: number analyzed (Participants) | 13 | 12 | 15
  Skin | 23.1 | 16.7 | 13.3
  Eyes: number analyzed (Participants) | 14 | 11 | 17
  Eyes | 35.7 | 36.4 | 23.5
  Mouth: number analyzed (Participants) | 13 | 11 | 11
  Mouth | 46.2 | 45.5 | 45.5
  Esophagus: number analyzed (Participants) | 2 | 0 | 4
  Esophagus | 50.0 |  | 25.0
  Upper GI tract: number analyzed (Participants) | 2 | 4 | 2
  Upper GI tract | 100.0 | 100.0 | 50.0
  Lower GI tract: number analyzed (Participants) | 1 | 2 | 1
  Lower GI tract | 0 | 100.0 | 0
  Liver: number analyzed (Participants) | 0 | 2 | 0
  Liver |  | 50.0 |
  Lungs: number analyzed (Participants) | 5 | 3 | 10
  Lungs | 0 | 0 | 30.0
  Joints and Fascia: number analyzed (Participants) | 11 | 11 | 12
  Joints and Fascia | 54.5 | 45.5 | 41.7

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from first dose of study drug to the death due to any reason. If there was no death, OS was censored by last visit, last long-term follow-up, or study cut-off date, whichever occurred first. Kaplan-Meier survival method was used for the analysis.
Time Frame: From first dose of study drug to date of death from any cause or data cut-off, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
months | NA [39.46 to NA] — Median and the corresponding 95% CI upper limits are not available because majority of the participants were still alive at the time of the final analysis. | NA [52.07 to NA] — Median and the corresponding 95% CI upper limits are not available because majority of the participants were still alive at the time of the final analysis. | NA [23.29 to NA] — Median and the corresponding 95% CI upper limits are not available because majority of the participants were still alive at the time of the final analysis.

13. Secondary Outcome: Time to Next Therapy (TTNT)
Description: The TTNT was defined as the time (in months) from first treatment to the time of new systemic cGVHD treatment. TTNT was censored by last response assessment or long term follow up assessment, whichever was earlier. Kaplan-Meier survival method was used for the analysis.
Time Frame: From time of first treatment to the time of new systemic cGVHD treatment or long term follow-up assessment, whichever occurred first (maximum duration: up to 64.2 months)
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
months | 15.2 [5.22 to NA] — 95% CI upper limit was not available due to the less number of participants with events (high percentage of censoring). | 9.8 [4.01 to 19.02] | 14.2 [2.66 to NA] — 95% CI upper limit was not available due to the less number of participants with events (high percentage of censoring).

14. Secondary Outcome: Change From Baseline in Overall Score on Lee cGvHD Symptom Scale at Specified Time Points
Description: Lee cGVHD symptom scale, a patient-reported symptom scale used to measure symptom burden and has 7 subscales (Skin, Eyes and Mouth, Breathing, Eating and Digestion, Muscles and Joints, Energy, and Mental and Emotional) with ratings as follows: 0-Not at all, 1-Slightly, 2-Moderately, 3-Quite a bit, 4-Extremely, with lower values representing better outcome. Score for each subscale was normalized to a score ranged from 0 to 100, where higher score=worse symptoms. An overall Lee cGvHD score was calculated as average of these 7 subscales and it ranged from 0 to 100, where a higher score = worse symptoms. EOT visit was performed within 3 days after the participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication.
Time Frame: Baseline, Day 1 of Cycles 2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18,19,20,21,22,23,24,25,26, 27,28,29,30,31,32,33,34,35,36,37, 38,39,40,41,42,43,44,45,46,47,48, 49, 50,51,52,53, 54,55, 56, 57,58,59,60,61,62,63,67 and EOT (i.e., anytime up to 64.2 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
score on a scale
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 8
  Cycle 2, Day 1 |  |  | -5.2 (6.3)
  Cycle 3, Day 1: number analyzed (Participants) | 16 | 12 | 16
  Cycle 3, Day 1 | -3.0 (8.5) | 0.5 (7.3) | -4.3 (8.2)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 9
  Cycle 4, Day 1 |  |  | -2.7 (8.2)
  Cycle 5, Day 1: number analyzed (Participants) | 13 | 10 | 12
  Cycle 5, Day 1 | -3.7 (11.0) | -3.7 (7.0) | -0.5 (10.8)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 12
  Cycle 6, Day 1 |  |  | -0.8 (9.3)
  Cycle 7, Day 1: number analyzed (Participants) | 10 | 9 | 12
  Cycle 7, Day 1 | -4.9 (8.4) | -2.2 (8.8) | -2.0 (12.3)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 2 | 11
  Cycle 8, Day 1 |  | -7.1 (10.1) | -2.9 (10.9)
  Cycle 9, Day 1: number analyzed (Participants) | 8 | 7 | 10
  Cycle 9, Day 1 | -3.7 (10.7) | -4.2 (5.5) | -3.6 (10.2)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 4 | 9
  Cycle 10, Day 1 |  | -2.7 (6.1) | -3.7 (9.9)
  Cycle 11, Day 1: number analyzed (Participants) | 7 | 6 | 9
  Cycle 11, Day 1 | -3.4 (11.5) | -5.5 (6.0) | -4.5 (6.1)
  Cycle 12, Day 1: number analyzed (Participants) | 2 | 5 | 8
  Cycle 12, Day 1 | -3.9 (8.1) | -7.6 (7.7) | -2.8 (6.0)
  Cycle 13, Day 1: number analyzed (Participants) | 6 | 5 | 7
  Cycle 13, Day 1 | -5.8 (14.7) | -5.9 (8.8) | -0.6 (7.1)
  Cycle 14, Day 1: number analyzed (Participants) | 5 | 5 | 7
  Cycle 14, Day 1 | -1.6 (17.1) | -5.0 (7.3) | -1.5 (7.7)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 4 | 7
  Cycle 15, Day 1 | -4.8 (15.8) | -6.8 (7.0) | -3.2 (8.2)
  Cycle 16, Day 1: number analyzed (Participants) | 5 | 3 | 4
  Cycle 16, Day 1 | -4.6 (16.1) | -6.9 (7.6) | 1.9 (7.9)
  Cycle 17, Day 1: number analyzed (Participants) | 5 | 3 | 5
  Cycle 17, Day 1 | -4.1 (17.2) | -10.1 (5.5) | 0.0 (12.5)
  Cycle 18, Day 1: number analyzed (Participants) | 5 | 3 | 3
  Cycle 18, Day 1 | -2.3 (17.6) | -11.5 (8.4) | -2.3 (7.8)
  Cycle 19, Day 1: number analyzed (Participants) | 5 | 3 | 4
  Cycle 19, Day 1 | -7.7 (19.6) | -9.9 (7.8) | -6.6 (9.9)
  Cycle 20, Day 1: number analyzed (Participants) | 5 | 3 | 3
  Cycle 20, Day 1 | -4.6 (22.0) | -9.0 (10.3) | -2.8 (5.6)
  Cycle 21, Day 1: number analyzed (Participants) | 5 | 3 | 4
  Cycle 21, Day 1 | -3.1 (19.1) | -7.5 (10.7) | -4.0 (7.9)
  Cycle 22, Day 1: number analyzed (Participants) | 5 | 2 | 3
  Cycle 22, Day 1 | -4.1 (18.9) | -14.5 (9.1) | -3.6 (5.0)
  Cycle 23, Day 1: number analyzed (Participants) | 5 | 2 | 4
  Cycle 23, Day 1 | -4.1 (19.1) | -11.6 (9.3) | -6.2 (7.7)
  Cycle 24, Day 1: number analyzed (Participants) | 4 | 1 | 2
  Cycle 24, Day 1 | -6.7 (21.0) | -18.7 | -5.6 (5.7)
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 25, Day 1 | 2.2 (18.8) | -12.4 (8.2) | -8.4 (3.4)
  Cycle 26, Day 1: number analyzed (Participants) | 3 | 0 | 1
  Cycle 26, Day 1 | 1.3 (14.3) |  | 0.2
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 27, Day 1 | -3.5 (25.3) | -13.2 (6.6) | -6.0 (9.6)
  Cycle 28, Day 1: number analyzed (Participants) | 3 | 0 | 1
  Cycle 28, Day 1 | 4.4 (13.4) |  | 2.6
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 29, Day 1 | -2.8 (23.7) | -11.0 (7.3) | -3.7 (13.0)
  Cycle 30, Day 1: number analyzed (Participants) | 2 | 0 | 0
  Cycle 30, Day 1 | 9.0 (7.5) |  |
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 31, Day 1 | -4.8 (27.9) | -15.6 (4.3) | -12.9
  Cycle 32, Day 1: number analyzed (Participants) | 2 | 0 | 0
  Cycle 32, Day 1 | 10.3 (6.9) |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 33, Day 1 | 0.5 (20.7) | -13.5 (9.0) | -12.9
  Cycle 34, Day 1: number analyzed (Participants) | 2 | 0 | 0
  Cycle 34, Day 1 | 13.5 (3.6) |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | -2.5 (23.3) | -11.0 (12.4) | -12.9
  Cycle 36, Day 1: number analyzed (Participants) | 2 | 0 | 0
  Cycle 36, Day 1 | 7.5 (6.4) |  |
  Cycle 37, Day 1: number analyzed (Participants) | 2 | 2 | 0
  Cycle 37, Day 1 | -5.3 (29.0) | -13.6 (8.1) |
  Cycle 38, Day 1: number analyzed (Participants) | 2 | 0 | 0
  Cycle 38, Day 1 | 9.1 (5.2) |  |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | -6.2 (25.9) | -14.3 (8.5) | -12.9
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | 2.7 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 41, Day 1 | -25.7 | -19.3 | -12.9
  Cycle 42, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 42, Day 1 | 4.6 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | -20.4 | -19.9 | -12.9
  Cycle 44, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 44, Day 1 | 4.3 |  |
  Cycle 45, Day 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 45, Day 1 |  |  | -12.3
  Cycle 46, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 46, Day 1 | 4.6 |  |
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 47, Day 1 | -6.8 | -16.8 | -12.9
  Cycle 48, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 48, Day 1 | 2.4 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 49, Day 1 |  | -15.4 | -14.3
  Cycle 50, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 50, Day 1 | 4.5 |  |
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 51, Day 1 | -12.0 |  | -12.9
  Cycle 52, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 52, Day 1 | 6.0 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | -19.2 |  |
  Cycle 54, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 54, Day 1 | 4.9 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | -16.8 |  |
  Cycle 56, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 56, Day 1 | 1.8 |  |
  Cycle 57, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 57, Day 1 | -17.6 |  |
  Cycle 58, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 58, Day 1 | 5.4 |  |
  Cycle 59, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 59, Day 1 | -12.7 |  |
  Cycle 60, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 60, Day 1 | 4.2 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | -19.3 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | 4.4 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | -18.0 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | -21.9 |  |
  EOT: number analyzed (Participants) | 10 | 8 | 10
  EOT | -4.3 (11.7) | -2.4 (10.9) | 2.5 (11.9)

15. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Each Specified Time Points
Description: FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline, Day 1 of Cycles 2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17,18,19,20,21,22,23,24,25,26,27, 29,30,31,32,33,34,35,36,37,38, 39,40,41,43, 47,48,49,51,52,53, 54, 55,56, 57,58,60,61,62,63,67, EOT (i.e., anytime up to 64.2 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
percent predicted FEV1
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 4
  Cycle 2, Day 1 |  |  | -4.8 (6.7)
  Cycle 3, Day 1: number analyzed (Participants) | 16 | 14 | 12
  Cycle 3, Day 1 | 1.1 (4.8) | -1.8 (7.1) | -1.5 (6.2)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 21
  Cycle 4, Day 1 |  |  | -0.2 (8.4)
  Cycle 5, Day 1: number analyzed (Participants) | 13 | 11 | 12
  Cycle 5, Day 1 | -3.3 (8.0) | -5.0 (6.5) | 0.5 (5.9)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 8
  Cycle 6, Day 1 |  |  | -0.9 (6.4)
  Cycle 7, Day 1: number analyzed (Participants) | 11 | 9 | 13
  Cycle 7, Day 1 | -3.5 (4.6) | -2.6 (9.4) | -0.9 (11.8)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 1 | 7
  Cycle 8, Day 1 |  | 1.0 | -1.1 (8.0)
  Cycle 9, Day 1: number analyzed (Participants) | 9 | 8 | 10
  Cycle 9, Day 1 | -1.7 (6.8) | -5.9 (11.7) | -3.0 (11.8)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 2 | 6
  Cycle 10, Day 1 |  | -6.0 (8.5) | 2.7 (3.9)
  Cycle 11, Day 1: number analyzed (Participants) | 7 | 6 | 8
  Cycle 11, Day 1 | -4.3 (5.2) | -4.0 (8.5) | -4.4 (15.8)
  Cycle 12, Day 1: number analyzed (Participants) | 1 | 1 | 7
  Cycle 12, Day 1 | -2.0 | -1.0 | 0.3 (3.6)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 4 | 8
  Cycle 13, Day 1 | -5.9 (9.3) | -2.5 (14.7) | -3.5 (13.2)
  Cycle 14, Day 1: number analyzed (Participants) | 1 | 1 | 7
  Cycle 14, Day 1 | 2.0 | 0.0 | -5.1 (9.1)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 3 | 8
  Cycle 15, Day 1 | -6.7 (11.7) | -2.3 (5.1) | -6.1 (12.6)
  Cycle 16, Day 1: number analyzed (Participants) | 1 | 2 | 4
  Cycle 16, Day 1 | 2.0 | -8.0 (15.6) | -4.5 (7.3)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 3 | 7
  Cycle 17, Day 1 | -5.3 (9.1) | -6.0 (7.2) | -7.9 (15.5)
  Cycle 18, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 18, Day 1 |  | -7.5 (10.6) | 4.0 (6.0)
  Cycle 19, Day 1: number analyzed (Participants) | 6 | 3 | 4
  Cycle 19, Day 1 | -5.2 (9.9) | -6.3 (5.5) | 0.5 (8.5)
  Cycle 20, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 20, Day 1 |  | -8.0 (7.1) | 4.0 (10.4)
  Cycle 21, Day 1: number analyzed (Participants) | 5 | 1 | 5
  Cycle 21, Day 1 | -7.4 (10.6) | 0.0 | -10.0 (19.8)
  Cycle 22, Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 22, Day 1 |  | -11.0 (1.4) | -6.0 (17.0)
  Cycle 23, Day 1: number analyzed (Participants) | 3 | 2 | 4
  Cycle 23, Day 1 | -4.3 (14.6) | -12.5 (4.9) | -4.8 (11.2)
  Cycle 24, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24, Day 1 | 2.0 | -18.0 | -19.0
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 25, Day 1 | -11.0 (15.6) | -12.5 (3.5) | -5.0 (11.4)
  Cycle 26, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 26, Day 1 | 0.0 |  |
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 27, Day 1 | -6.5 (13.4) | -17.0 (9.9) | -10.0 (17.0)
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 29, Day 1 | -0.5 (9.2) | 17.0 (11.3) | 0.0 (1.4)
  Cycle 30, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 30, Day 1 | 3.0 |  |
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 31, Day 1 | -3.5 (12.0) | -19.5 (10.6) | -4.0
  Cycle 32, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 32, Day 1 | 1.0 |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 2 | 0
  Cycle 33, Day 1 | 5.0 (5.7) | -1.0 (33.9) |
  Cycle 34, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 34, Day 1 | 2.0 |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | 5.0 (0.0) | -2.5 (30.4) | -4.0
  Cycle 36, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 36, Day 1 | 3.0 |  | 5.0
  Cycle 37, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 37, Day 1 | -1.0 | -22.0 |
  Cycle 38, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 38, Day 1 | 1.0 |  |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | 10.0 (2.8) | -23.0 (11.3) | -5.0
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | -1.0 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 41, Day 1 | 15.0 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | 16.0 | -21.0 | -7.0
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 47, Day 1 | 5.0 |  | -5.0
  Cycle 48, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 48, Day 1 | 3.0 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 49, Day 1 | 8.0 |  | -2.0
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 51, Day 1 | 8.0 |  |
  Cycle 52, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 52, Day 1 | 0.0 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | 9.0 |  |
  Cycle 54, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 54, Day 1 | 4.0 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | 13.0 |  |
  Cycle 56, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 56, Day 1 | 4.0 |  |
  Cycle 57, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 57, Day 1 | 13.0 |  |
  Cycle 58, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 58, Day 1 | 5.0 |  |
  Cycle 60, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 60, Day 1 | 4.0 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | 10.0 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | 2.0 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | 13.0 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | 14.0 |  |
  EOT: number analyzed (Participants) | 12 | 10 | 9
  EOT | -1.4 (9.0) | -10.1 (15.7) | -7.4 (14.9)

16. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Each Specified Time Points
Description: FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline, Day 1 of Cycles 2, 3,4, 5,6,7,8,9,10,11,12,13, 14,15,16,17,18,19,20,21,22,23,24,25,26, 27,29,30,31,32,33,34,35,36,37,38,39,40,41,43,47, 48,49, 51,52,53,54, 55, 56,57,58,60,61, 62, 63,67, EOT (i.e., anytime up to 64.2 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
percent predicted FVC
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 4
  Cycle 2, Day 1 |  |  | -5.5 (9.9)
  Cycle 3, Day 1: number analyzed (Participants) | 16 | 14 | 12
  Cycle 3, Day 1 | 0.5 (3.8) | -2.4 (6.0) | -3.0 (6.7)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 6
  Cycle 4, Day 1 |  |  | -0.2 (8.6)
  Cycle 5, Day 1: number analyzed (Participants) | 13 | 11 | 12
  Cycle 5, Day 1 | -0.5 (7.1) | -4.3 (5.2) | 1.6 (6.3)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 8
  Cycle 6, Day 1 |  |  | 0.8 (9.5)
  Cycle 7, Day 1: number analyzed (Participants) | 11 | 9 | 13
  Cycle 7, Day 1 | -2.9 (5.2) | -1.3 (6.4) | 2.3 (9.7)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 1 | 7
  Cycle 8, Day 1 |  | 2.0 | 0.4 (8.9)
  Cycle 9, Day 1: number analyzed (Participants) | 9 | 8 | 10
  Cycle 9, Day 1 | 0.4 (5.1) | -2.9 (5.5) | -0.8 (9.5)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 2 | 6
  Cycle 10, Day 1 |  | -5.0 (8.5) | 4.7 (4.9)
  Cycle 11, Day 1: number analyzed (Participants) | 7 | 6 | 8
  Cycle 11, Day 1 | -1.1 (7.3) | -2.7 (5.6) | -4.4 (12.0)
  Cycle 12, Day 1: number analyzed (Participants) | 1 | 1 | 7
  Cycle 12, Day 1 | 2.0 | 1.0 | 0.7 (5.8)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 4 | 8
  Cycle 13, Day 1 | -2.4 (7.9) | -3.3 (15.4) | -4.9 (9.8)
  Cycle 14, Day 1: number analyzed (Participants) | 1 | 1 | 7
  Cycle 14, Day 1 | 11.0 | 2.0 | -2.7 (7.1)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 3 | 8
  Cycle 15, Day 1 | -3.7 (10.4) | -3.3 (5.5) | -4.8 (11.5)
  Cycle 16, Day 1: number analyzed (Participants) | 1 | 2 | 4
  Cycle 16, Day 1 | 16.0 | -6.0 (19.8) | -6.5 (6.5)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 3 | 7
  Cycle 17, Day 1 | -3.2 (6.3) | -3.0 (11.8) | -5.6 (12.8)
  Cycle 18, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 18, Day 1 |  | -7.5 (9.2) | 4.0 (4.0)
  Cycle 19, Day 1: number analyzed (Participants) | 6 | 3 | 4
  Cycle 19, Day 1 | -2.3 (6.8) | -5.3 (4.7) | 0.8 (5.1)
  Cycle 20, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 20, Day 1 |  | -10.5 (2.1) | -2.0 (5.6)
  Cycle 21, Day 1: number analyzed (Participants) | 5 | 1 | 5
  Cycle 21, Day 1 | -3.2 (8.1) | -3.0 | -6.6 (17.0)
  Cycle 22, Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 22, Day 1 |  | -11.0 (0.0) | -6.0 (8.5)
  Cycle 23, Day 1: number analyzed (Participants) | 3 | 2 | 4
  Cycle 23, Day 1 | 0.0 (12.3) | -11.0 (2.8) | -1.8 (10.6)
  Cycle 24, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24, Day 1 | 4.0 | -13.0 | -15.0
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 25, Day 1 | -7.0 (11.3) | -10.5 (3.5) | -1.3 (11.7)
  Cycle 26, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 26, Day 1 | 4.0 |  |
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 27, Day 1 | -2.0 (4.2) | -18.0 (12.7) | -4.0 (21.2)
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 1 | 2
  Cycle 29, Day 1 | 2.5 (4.9) | -11.0 | 6.0 (1.4)
  Cycle 30, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 30, Day 1 | 4.0 |  |
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 31, Day 1 | 1.5 (3.5) | -15.5 (7.8) | -4.0
  Cycle 32, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 32, Day 1 | 2.0 |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 2 | 0
  Cycle 33, Day 1 | 11.0 (0.0) | -17.5 (7.8) |
  Cycle 34, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 34, Day 1 | 6.0 |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | 11.0 (5.7) | -15.0 (11.3) | -3.0
  Cycle 36, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 36, Day 1 | 5.0 |  | 2.0
  Cycle 37, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 37, Day 1 | 7.0 | -24.0 |
  Cycle 38, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 38, Day 1 | 2.0 |  |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | 12.5 (0.7) | -20.5 (12.0) | -1.0
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | 3.0 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 41, Day 1 | 15.0 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | 17.0 | -18.0 | -4.0
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 47, Day 1 | 5.0 |  | -2.0
  Cycle 48, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 48, Day 1 | 5.0 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 49, Day 1 | 6.0 |  | 2.0
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 51, Day 1 | 9.0 |  |
  Cycle 52, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 52, Day 1 | 3.0 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | 8.0 |  |
  Cycle 54, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 54, Day 1 | 5.0 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | 13.0 |  |
  Cycle 56, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 56, Day 1 | 7.0 |  |
  Cycle 57, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 57, Day 1 | 14.0 |  |
  Cycle 58, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 58, Day 1 | 7.0 |  |
  Cycle 60, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 60, Day 1 | 8.0 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | 12.0 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | 5.0 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | 12.0 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | 14.0 |  |
  EOT: number analyzed (Participants) | 12 | 10 | 9
  EOT | -2.5 (10.3) | -8.4 (9.2) | -7.8 (14.7)

17. Secondary Outcome: Change From Baseline in Percent Predicted Hemoglobin (HGB) Corrected Diffusing Capacity of Lung for Carbon Monoxide (DLco) at Each Specified Time Points
Description: DLco is a measurement of the ability of the lungs to transfer gases from the air to the blood. Change from baseline in diffusing capacity of the lung for carbon monoxide (percent predicted hemoglobin level corrected) was reported for this measure. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline, Day 1 of Cycles 2,3,4,5,6,7,8,9,10,11,12,13, 14,15,16,17,18,19,20,21,22,23,24,25,26,27, 29,31,32,33,34,35,36,37,39,40,41,43,47,49,51,53,55, 61, 62, 63, 67, EOT (i.e., anytime up to 64.2 Months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent Predicted HGB Corrected DLco
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Percent Predicted HGB Corrected DLco
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 4
  Cycle 2, Day 1 |  |  | -5.243 (9.830)
  Cycle 3, Day 1: number analyzed (Participants) | 14 | 14 | 9
  Cycle 3, Day 1 | 4.545 (22.991) | -0.638 (7.059) | -3.928 (9.492)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 5
  Cycle 4, Day 1 |  |  | 0.278 (9.683)
  Cycle 5, Day 1: number analyzed (Participants) | 12 | 12 | 9
  Cycle 5, Day 1 | 4.635 (23.989) | -4.462 (23.621) | -4.111 (9.138)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 7
  Cycle 6, Day 1 |  |  | -3.143 (10.385)
  Cycle 7, Day 1: number analyzed (Participants) | 10 | 8 | 7
  Cycle 7, Day 1 | 1.521 (19.836) | 6.184 (9.436) | -4.275 (11.464)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 1 | 6
  Cycle 8, Day 1 |  | 3.554 | -3.787 (11.983)
  Cycle 9, Day 1: number analyzed (Participants) | 9 | 8 | 8
  Cycle 9, Day 1 | -4.514 (7.401) | 2.570 (8.902) | -2.540 (11.897)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 2 | 5
  Cycle 10, Day 1 |  | 4.343 (3.144) | 1.328 (8.887)
  Cycle 11, Day 1: number analyzed (Participants) | 6 | 6 | 7
  Cycle 11, Day 1 | -0.625 (7.262) | 6.582 (10.695) | -2.720 (10.920)
  Cycle 12, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 12, Day 1 | 0.531 | 4.076 | -1.378 (6.364)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 4 | 7
  Cycle 13, Day 1 | -5.548 (12.175) | 1.882 (7.522) | 2.091 (13.290)
  Cycle 14, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 14, Day 1 | 12.916 | 0.358 | 0.309 (11.651)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 3 | 7
  Cycle 15, Day 1 | 0.228 (15.731) | 1.125 (5.927) | -5.309 (11.514)
  Cycle 16, Day 1: number analyzed (Participants) | 1 | 2 | 4
  Cycle 16, Day 1 | 48.465 | -6.618 (15.443) | -6.840 (15.053)
  Cycle 17, Day 1: number analyzed (Participants) | 6 | 3 | 6
  Cycle 17, Day 1 | -1.018 (9.226) | 8.458 (6.229) | -10.865 (13.346)
  Cycle 18, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 18, Day 1 |  | 15.543 (11.753) | -3.174 (3.106)
  Cycle 19, Day 1: number analyzed (Participants) | 6 | 3 | 3
  Cycle 19, Day 1 | -2.293 (5.763) | 1.824 (8.539) | -2.020 (2.436)
  Cycle 20, Day 1: number analyzed (Participants) | 0 | 1 | 3
  Cycle 20, Day 1 |  | -14.692 | -13.517 (5.936)
  Cycle 21, Day 1: number analyzed (Participants) | 5 | 1 | 4
  Cycle 21, Day 1 | -2.778 (8.187) | -10.661 | -12.354 (12.800)
  Cycle 22, Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 22, Day 1 |  | 3.347 (3.560) | -17.222 (16.947)
  Cycle 23, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 23, Day 1 | 0.354 (1.844) | -15.184 (20.181) | -2.219 (10.614)
  Cycle 24, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24, Day 1 | 6.945 | -18.095 | -11.430
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 25, Day 1 | -4.461 (19.865) | 6.289 (2.469) | -13.392
  Cycle 26, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 26, Day 1 | 4.715 |  |
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 27, Day 1 | -8.047 (24.788) | -9.914 (15.387) | -11.154
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 29, Day 1 | -6.701 (1.671) | -18.814 (24.960) | 8.613
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 31, Day 1 | 2.343 (20.988) | -0.800 (17.528) | 10.833
  Cycle 32, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 32, Day 1 | 5.586 |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 2 | 0
  Cycle 33, Day 1 | 9.901 (9.954) | -5.962 (10.550) |
  Cycle 34, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 34, Day 1 | 4.863 |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | 13.867 (1.309) | -0.426 (6.677) | 5.088
  Cycle 36, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 36, Day 1 | 4.166 |  | 10.372
  Cycle 37, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 37, Day 1 | 9.306 | -19.228 |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | 14.754 (0.649) | -6.813 (12.810) | 5.902
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | 5.586 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 41, Day 1 | 22.884 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | 15.213 | 8.775 | 16.351
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 47, Day 1 | 9.660 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 49, Day 1 | -3.599 |  |
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 51, Day 1 | 11.734 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | 10.292 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | 16.550 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | 17.682 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | 4.170 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | 26.215 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | 41.384 |  |
  EOT: number analyzed (Participants) | 9 | 6 | 7
  EOT | -1.962 (11.426) | 0.985 (5.919) | -10.371 (14.208)

18. Secondary Outcome: Change From Baseline in Percent Predicted Total Lung Capacity (TLC) at Each Specified Time Points
Description: TLC is the volume of air in the lungs upon the maximum effort of inspiration. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline, Day 1 of Cycles 2,3, 4, 5,6,7, 8, 9, 10,11,12,13, 14, 15, 16, 17, 18, 19, 20,21, 22,23,24, 25, 26, 27,29, 30, 31,32, 33, 34, 35,36, 37, 38,39, 40,41,43,47, 48, 49,51,52,53, 54,55,56,57,58, 60,61,62, 63, 67, EOT (i.e., anytime up to 64.2 Months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent Predicted TLC
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
Percent Predicted TLC
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 4
  Cycle 2, Day 1 |  |  | -9.0 (13.4)
  Cycle 3, Day 1: number analyzed (Participants) | 14 | 12 | 12
  Cycle 3, Day 1 | 1.6 (11.9) | 1.9 (8.5) | -0.6 (14.8)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 6
  Cycle 4, Day 1 |  |  | 3.3 (14.0)
  Cycle 5, Day 1: number analyzed (Participants) | 13 | 9 | 10
  Cycle 5, Day 1 | -2.6 (16.8) | -7.2 (10.5) | -1.7 (11.2)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 7
  Cycle 6, Day 1 |  |  | -4.4 (11.6)
  Cycle 7, Day 1: number analyzed (Participants) | 11 | 7 | 12
  Cycle 7, Day 1 | -3.7 (6.6) | -4.4 (6.3) | -2.6 (13.4)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 1 | 6
  Cycle 8, Day 1 |  | -5.0 | -0.2 (12.9)
  Cycle 9, Day 1: number analyzed (Participants) | 9 | 8 | 10
  Cycle 9, Day 1 | -2.9 (6.1) | -6.0 (8.5) | -0.9 (15.8)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 2 | 5
  Cycle 10, Day 1 |  | -18.5 (6.4) | 3.6 (14.7)
  Cycle 11, Day 1: number analyzed (Participants) | 7 | 6 | 8
  Cycle 11, Day 1 | 0.7 (4.3) | -5.2 (11.2) | -3.0 (19.7)
  Cycle 12, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 12, Day 1 | -9.0 | 0.0 | -8.0 (14.2)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 4 | 8
  Cycle 13, Day 1 | -0.3 (7.1) | -10.3 (18.7) | -3.3 (17.6)
  Cycle 14, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 14, Day 1 | 23.0 | -7.0 | -5.8 (16.5)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 3 | 7
  Cycle 15, Day 1 | -2.8 (10.8) | -1.0 (5.6) | -7.0 (12.0)
  Cycle 16, Day 1: number analyzed (Participants) | 1 | 2 | 4
  Cycle 16, Day 1 | -3.0 | -14.0 (12.7) | -15.5 (9.5)
  Cycle 17, Day 1: number analyzed (Participants) | 5 | 3 | 7
  Cycle 17, Day 1 | -3.0 (6.2) | -17.0 (11.4) | -18.1 (15.6)
  Cycle 18, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 18, Day 1 |  | -16.0 (8.5) | 0.0 (13.9)
  Cycle 19, Day 1: number analyzed (Participants) | 5 | 3 | 4
  Cycle 19, Day 1 | -4.6 (6.1) | -7.7 (10.5) | -7.0 (5.4)
  Cycle 20, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 20, Day 1 |  | -9.5 (16.3) | -9.3 (15.4)
  Cycle 21, Day 1: number analyzed (Participants) | 3 | 1 | 5
  Cycle 21, Day 1 | 0.3 (9.3) | -18.0 | -14.4 (24.0)
  Cycle 22, Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 22, Day 1 |  | -18.5 (6.4) | -21.0 (14.1)
  Cycle 23, Day 1: number analyzed (Participants) | 3 | 2 | 4
  Cycle 23, Day 1 | 0.0 (8.7) | -21.0 (19.8) | -2.8 (18.8)
  Cycle 24, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24, Day 1 | 0.0 | -15.0 | -34.0
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 25, Day 1 | -3.0 (7.1) | -19.5 (13.4) | -6.3 (24.1)
  Cycle 26, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 26, Day 1 | 0.0 |  |
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 27, Day 1 | 5.5 (16.3) | -24.0 (12.7) | -14.5 (24.7)
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 29, Day 1 | -1.0 (17.0) | -27.5 (21.9) | 12.0 (14.1)
  Cycle 30, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 30, Day 1 | 7.0 |  |
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 1 | 1
  Cycle 31, Day 1 | 7.5 (17.7) | -36.0 | 17.0
  Cycle 32, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 32, Day 1 | 1.0 |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 1 | 0
  Cycle 33, Day 1 | 14.0 (11.3) | -39.0 |
  Cycle 34, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 34, Day 1 | 2.0 |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | 10.5 (7.8) | -23.5 (16.3) | 13.0
  Cycle 36, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 36, Day 1 | 6.0 |  | -6.0
  Cycle 37, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 37, Day 1 | -7.0 | -41.0 |
  Cycle 38, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 38, Day 1 | 2.0 |  |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | 24.0 (28.3) | -30.0 (21.2) | 23.0
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | 0.0 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 41, Day 1 | 38.0 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | 33.0 | -16.0 | 21.0
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 47, Day 1 | 19.0 |  | 25.0
  Cycle 48, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 48, Day 1 | -13.0 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 49, Day 1 | 5.0 |  | 1.0
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 51, Day 1 | 15.0 |  |
  Cycle 52, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 52, Day 1 | 1.0 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | 15.0 |  |
  Cycle 54, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 54, Day 1 | 4.0 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | 29.0 |  |
  Cycle 56, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 56, Day 1 | 9.0 |  |
  Cycle 57, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 57, Day 1 | 18.0 |  |
  Cycle 58, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 58, Day 1 | 5.0 |  |
  Cycle 60, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 60, Day 1 | -3.0 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | 5.0 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | -1.0 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | 12.0 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | 12.0 |  |
  EOT: number analyzed (Participants) | 10 | 7 | 8
  EOT | 5.2 (27.5) | -2.4 (15.0) | -12.6 (20.1)

19. Secondary Outcome: Change From Baseline in Percent Predicted Residual Volume (RV) at Each Specified Time Points
Description: RV is the volume of air remaining in the lungs after maximum forceful expiration. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 3 days after the participant's last dose of study drug.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4,5, 6,7, 8, 9, 10, 11,12, 13, 14,15, 16,17, 18, 19,20, 21,22,23, 24, 25, 26,27, 29, 30, 31, 32, 33,34, 35,36, 37,38, 39, 40,41, 43,47, 48, 49,51,52,53, 54, 55,56,57, 58,60,61,62,63,67, EOT (i.e., anytime up to 64.2 Months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent predicted RV
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
percent predicted RV
  Cycle 2, Day 1: number analyzed (Participants) | 0 | 0 | 4
  Cycle 2, Day 1 |  |  | -18.0 (30.1)
  Cycle 3, Day 1: number analyzed (Participants) | 14 | 12 | 12
  Cycle 3, Day 1 | 0.2 (22.2) | -4.6 (18.8) | 9.0 (34.4)
  Cycle 4, Day 1: number analyzed (Participants) | 0 | 0 | 6
  Cycle 4, Day 1 |  |  | 17.8 (29.0)
  Cycle 5, Day 1: number analyzed (Participants) | 13 | 11 | 10
  Cycle 5, Day 1 | 5.2 (24.5) | -11.5 (26.9) | -3.7 (29.8)
  Cycle 6, Day 1: number analyzed (Participants) | 0 | 0 | 7
  Cycle 6, Day 1 |  |  | -10.9 (37.5)
  Cycle 7, Day 1: number analyzed (Participants) | 11 | 8 | 12
  Cycle 7, Day 1 | 4.9 (29.1) | -9.9 (17.1) | -7.5 (33.0)
  Cycle 8, Day 1: number analyzed (Participants) | 0 | 1 | 6
  Cycle 8, Day 1 |  | -28.0 | 2.5 (39.7)
  Cycle 9, Day 1: number analyzed (Participants) | 9 | 8 | 10
  Cycle 9, Day 1 | 6.4 (27.4) | -19.9 (24.3) | 0.1 (35.6)
  Cycle 10, Day 1: number analyzed (Participants) | 0 | 2 | 5
  Cycle 10, Day 1 |  | -47.5 (0.7) | 1.4 (38.2)
  Cycle 11, Day 1: number analyzed (Participants) | 7 | 6 | 8
  Cycle 11, Day 1 | 22.1 (29.6) | -10.5 (28.3) | 5.4 (38.0)
  Cycle 12, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 12, Day 1 | -28.0 | -5.0 | -22.2 (49.9)
  Cycle 13, Day 1: number analyzed (Participants) | 7 | 4 | 8
  Cycle 13, Day 1 | 20.3 (19.9) | -27.0 (35.6) | 0.3 (32.6)
  Cycle 14, Day 1: number analyzed (Participants) | 1 | 1 | 6
  Cycle 14, Day 1 | 78.0 | -31.0 | -6.5 (36.3)
  Cycle 15, Day 1: number analyzed (Participants) | 6 | 3 | 7
  Cycle 15, Day 1 | 20.3 (27.4) | -0.7 (18.1) | -16.7 (22.3)
  Cycle 16, Day 1: number analyzed (Participants) | 1 | 2 | 4
  Cycle 16, Day 1 | 0.0 | -36.5 (13.4) | -27.5 (31.9)
  Cycle 17, Day 1: number analyzed (Participants) | 5 | 3 | 7
  Cycle 17, Day 1 | 13.6 (27.8) | -47.3 (25.1) | -39.1 (26.2)
  Cycle 18, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 18, Day 1 |  | -42.0 (0.0) | -7.3 (33.7)
  Cycle 19, Day 1: number analyzed (Participants) | 5 | 3 | 4
  Cycle 19, Day 1 | 5.4 (28.7) | -19.7 (18.0) | -23.5 (18.7)
  Cycle 20, Day 1: number analyzed (Participants) | 0 | 2 | 3
  Cycle 20, Day 1 |  | -7.5 (37.5) | -22.0 (44.3)
  Cycle 21, Day 1: number analyzed (Participants) | 3 | 1 | 5
  Cycle 21, Day 1 | 8.3 (10.0) | -44.0 | -30.2 (51.2)
  Cycle 22, Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 22, Day 1 |  | -33.0 (19.8) | -41.0 (46.7)
  Cycle 23, Day 1: number analyzed (Participants) | 3 | 1 | 4
  Cycle 23, Day 1 | 0.3 (5.1) | -72.0 | 1.5 (44.8)
  Cycle 24, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 24, Day 1 | -4.0 | -17.0 | -78.0
  Cycle 25, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 25, Day 1 | 1.0 (9.9) | -34.0 (31.1) | -23.3 (56.0)
  Cycle 26, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 26, Day 1 | -3.0 |  |
  Cycle 27, Day 1: number analyzed (Participants) | 2 | 2 | 2
  Cycle 27, Day 1 | 19.5 (41.7) | -39.5 (20.5) | -41.0 (28.3)
  Cycle 29, Day 1: number analyzed (Participants) | 2 | 1 | 2
  Cycle 29, Day 1 | -13.0 (42.4) | -13.0 | 17.5 (40.3)
  Cycle 30, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 30, Day 1 | 21.0 |  |
  Cycle 31, Day 1: number analyzed (Participants) | 2 | 1 | 1
  Cycle 31, Day 1 | 15.0 (43.8) | -93.0 | 61.0
  Cycle 32, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 32, Day 1 | 5.0 |  |
  Cycle 33, Day 1: number analyzed (Participants) | 2 | 1 | 0
  Cycle 33, Day 1 | 14.5 (36.1) | -70.0 |
  Cycle 34, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 34, Day 1 | -1.0 |  |
  Cycle 35, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 35, Day 1 | 3.5 (36.1) | -34.5 (33.2) | 47.0
  Cycle 36, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 36, Day 1 | 17.0 |  | -20.0
  Cycle 37, Day 1: number analyzed (Participants) | 1 | 1 | 0
  Cycle 37, Day 1 | -54.0 | -70.0 |
  Cycle 38, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 38, Day 1 | 8.0 |  |
  Cycle 39, Day 1: number analyzed (Participants) | 2 | 2 | 1
  Cycle 39, Day 1 | 43.0 (89.1) | -43.0 (42.4) | 81.0
  Cycle 40, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 40, Day 1 | -1.0 |  |
  Cycle 41, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 41, Day 1 | 80.0 |  |
  Cycle 43, Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 43, Day 1 | 58.0 | -26.0 | 75.0
  Cycle 47, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 47, Day 1 | 42.0 |  | 87.0
  Cycle 48, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 48, Day 1 | -50.0 |  |
  Cycle 49, Day 1: number analyzed (Participants) | 1 | 0 | 1
  Cycle 49, Day 1 | -14.0 |  | -5.0
  Cycle 51, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 51, Day 1 | 22.0 |  |
  Cycle 52, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 52, Day 1 | -4.0 |  |
  Cycle 53, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 53, Day 1 | 22.0 |  |
  Cycle 54, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 54, Day 1 | 4.0 |  |
  Cycle 55, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 55, Day 1 | 53.0 |  |
  Cycle 56, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 56, Day 1 | 17.0 |  |
  Cycle 57, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 57, Day 1 | 18.0 |  |
  Cycle 58, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 58, Day 1 | 4.0 |  |
  Cycle 60, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 60, Day 1 | -20.0 |  |
  Cycle 61, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 61, Day 1 | -18.0 |  |
  Cycle 62, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 62, Day 1 | -8.0 |  |
  Cycle 63, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 63, Day 1 | 6.0 |  |
  Cycle 67, Day 1: number analyzed (Participants) | 1 | 0 | 0
  Cycle 67, Day 1 | 2.0 |  |
  EOT: number analyzed (Participants) | 11 | 8 | 8
  EOT | 6.3 (24.3) | 10.6 (34.9) | -18.5 (32.6)

20. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Belumosudil and Its Metabolites (KD025m1 and KD025m2)
Description: Cmax was the maximum observed plasma concentration, obtained by a non-compartmental analysis. Cmax data for Belumosudil and its metabolites KD025m1 and KD025m2 are reported in this outcome measure.
Time Frame: Cycles 1 and 2: pre-dose (0 hour), 1, 2, 3, 4, 5, and 6 hours post-dose on Day 1
Population: Analysis was performed on PK population which included all participants who received at least one dose of study drug and had at least 1 post-dose PK sample drawn. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
nanograms per milliliter
  Belumosudil: Cycle 1 Day 1: number analyzed (Participants) | 16 | 16 | 21
  Belumosudil: Cycle 1 Day 1 | 2500 (60.1) | 1400 (98.5) | 2960 (69.7)
  Belumosudil: Cycle 2 Day 1: number analyzed (Participants) | 16 | 14 | 16
  Belumosudil: Cycle 2 Day 1 | 2020 (101) | 1890 (120) | 3270 (63.0)
  KD025m1: Cycle 1 Day 1: number analyzed (Participants) | 6 | 6 | 14
  KD025m1: Cycle 1 Day 1 | 44.4 (67.9) | 34.8 (58.8) | 63.9 (59.4)
  KD025m1: Cycle 2 Day 1: number analyzed (Participants) | 7 | 5 | 11
  KD025m1: Cycle 2 Day 1 | 36.2 (43.0) | 45.0 (38.6) | 55.8 (82.1)
  KD025m2: Cycle 1 Day 1: number analyzed (Participants) | 15 | 14 | 17
  KD025m2: Cycle 1 Day 1 | 208 (93.1) | 99.2 (112) | 388 (82.3)
  KD025m2: Cycle 2 Day 1: number analyzed (Participants) | 15 | 13 | 16
  KD025m2: Cycle 2 Day 1 | 158 (150) | 145 (147) | 265 (154)

21. Secondary Outcome: Pharmacokinetics: Time of the Maximum Observed Plasma Concentration (Tmax) of Belumosudil and Its Metabolites (KD025m1 and KD025m2)
Description: Tmax was defined as time to reach maximum observed plasma concentration, obtained by a non-compartmental analysis. Tmax data for Belumosudil and its metabolites KD025m1 and KD025m2 are reported in this outcome measure.
Time Frame: Cycles 1 and 2: pre-dose (0 hour), 1, 2, 3, 4, 5, and 6 hours post-dose on Day 1
Population: Analysis was performed on PK population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
hours
  Belumosudil: Cycle 1 Day 1: number analyzed (Participants) | 16 | 16 | 21
  Belumosudil: Cycle 1 Day 1 | 2.12 [0.98 to 5.00] | 3.43 [1.97 to 6.00] | 3.03 [1.85 to 6.00]
  Belumosudil: Cycle 2 Day 1: number analyzed (Participants) | 16 | 14 | 16
  Belumosudil: Cycle 2 Day 1 | 2.53 [0 to 4.87] | 2.47 [0 to 5.83] | 2.66 [1.00 to 6.02]
  KD025m1: Cycle 1 Day 1: number analyzed (Participants) | 6 | 6 | 14
  KD025m1: Cycle 1 Day 1 | 2.50 [1.00 to 3.98] | 1.75 [1.08 to 5.95] | 1.98 [0.90 to 4.95]
  KD025m1: Cycle 2 Day 1: number analyzed (Participants) | 7 | 5 | 11
  KD025m1: Cycle 2 Day 1 | 2.98 [1.17 to 3.03] | 2.05 [1.08 to 5.83] | 2.17 [1.00 to 4.03]
  KD025m2: Cycle 1 Day 1: number analyzed (Participants) | 15 | 14 | 17
  KD025m2: Cycle 1 Day 1 | 2.82 [1.93 to 5.00] | 3.00 [2.00 to 6.00] | 2.98 [1.85 to 6.00]
  KD025m2: Cycle 2 Day 1: number analyzed (Participants) | 15 | 13 | 16
  KD025m2: Cycle 2 Day 1 | 2.98 [0 to 3.93] | 2.00 [1.05 to 5.07] | 3.03 [1.98 to 6.02]

22. Secondary Outcome: Pharmacokinetics: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to 6 Hours Post-dose (AUC0-6hr) of Belumosudil and Its Metabolites (KD025m1 and KD025m2)
Description: AUC0-6hr was defined as area under the plasma concentration versus time curve from time 0 to 6 hours post-dose, obtained by a non-compartmental analysis from the concentration-time data. AUC0-6hr data for Belumosudil and its metabolites KD025m1 and KD025m2 are reported in this outcome measure.
Time Frame: Cycles 1 and 2: pre-dose (0 hour), 1, 2, 3, 4, 5, and 6 hours post-dose on Day 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter
Arm/Group | Cohort 1: Belumosudil 200 mg QD | Cohort 2: Belumosudil 200 mg BID | Cohort 3: Belumosudil 400 mg QD
Number analyzed (Participants) | 17 | 16 | 21
hours*nanograms per milliliter
  Belumosudil: Cycle 1 Day 1: number analyzed (Participants) | 16 | 16 | 21
  Belumosudil: Cycle 1 Day 1 | 8350 (60.3) | 4960 (108) | 11500 (97.3)
  Belumosudil: Cycle 2 Day 1: number analyzed (Participants) | 16 | 14 | 16
  Belumosudil: Cycle 2 Day 1 | 7090 (95.9) | 7190 (115) | 12000 (68.8)
  KD025m1: Cycle 1 Day 1: number analyzed (Participants) | 6 | 6 | 14
  KD025m1: Cycle 1 Day 1 | 140 (72.3) | 114 (60.8) | 216 (61.9)
  KD025m1: Cycle 2 Day 1: number analyzed (Participants) | 7 | 5 | 11
  KD025m1: Cycle 2 Day 1 | 123 (38.2) | 160 (31.3) | 178 (72.9)
  KD025m2: Cycle 1 Day 1: number analyzed (Participants) | 15 | 14 | 17
  KD025m2: Cycle 1 Day 1 | 565 (90.8) | 282 (125) | 1150 (97.1)
  KD025m2: Cycle 2 Day 1: number analyzed (Participants) | 15 | 13 | 16
  KD025m2: Cycle 2 Day 1 | 471 (145) | 513 (122) | 923 (144)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after the last dose of study drug (maximum duration: up to 64.2 months)
Description: Analysis was performed on the safety population. Disease progression related death was not reported as AE.
Groups:
- Cohort 1 200 mg QD: Participants received belumosudil 200 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 64.2 months).
- Cohort 2 200 mg BID: Participants received belumosudil 200 mg orally BID in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 45.9 months).
- Cohort 3 400 mg QD: Participants received belumosudil 400 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first (maximum duration: 49.2 months).
Arm/Group | Cohort 1 200 mg QD | Cohort 2 200 mg BID | Cohort 3 400 mg QD
All-Cause Mortality (participants affected / at risk) | 5/17 | 5/16 | 9/21
Serious Adverse Events (participants affected / at risk) | 5/17 | 6/16 | 13/21
Other Adverse Events (participants affected / at risk) | 17/17 | 16/16 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 200 mg QD (N=17) | Cohort 2 200 mg BID (N=16) | Cohort 3 400 mg QD (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in lung (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Citrobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 3 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Respirovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipomatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy of partner (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 200 mg QD (N=17) | Cohort 2 200 mg BID (N=16) | Cohort 3 400 mg QD (N=21)
Anaemia (Blood and lymphatic system disorders) | 5 (14) | 4 (8) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Hypogonadism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 1 (2) | 3 (4)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 2 (3) | 4 (4) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (4) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (4) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 5 (10) | 7 (11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (3)
Enamel anomaly (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (10) | 4 (6) | 9 (12)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4) | 3 (3) | 4 (4)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (7) | 3 (7) | 10 (14)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 4 (5) | 6 (6)
Pain (General disorders) | 3 (3) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (3) | 3 (6) | 3 (3)
Contrast media allergy (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Corneal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (2) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 3 (3) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (4) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (16) | 9 (13) | 7 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (4)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (12) | 3 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (8) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bronchoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (9) | 4 (4) | 0 (0)
Glucose urine present (Investigations) | 2 (3) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (4)
Weight increased (Investigations) | 3 (9) | 1 (2) | 1 (4)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2) | 3 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (6) | 1 (2) | 3 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 4 (5)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (4) | 2 (2)
Epidural lipomatosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 6 (8)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (3) | 1 (2) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (3) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (4) | 2 (2) | 2 (6)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (4) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (7) | 1 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 2 (5) | 4 (6)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT02841995/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT02841995/SAP_001.pdf